CLINICAL TRIAL: NCT05814315
Title: Opioid Support and Risk Reduction Online Platform
Brief Title: Harnessing Online Peer Education Opioid Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElevateU (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ElevateU
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Medication Compliance; Pain
MeSH Terms: conditions — Medication Adherence; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE Intervention (Experimental): These participants will have peer support and online support groups.
  Interventions: Behavioral: HOPE Intervention
- Control (No Intervention): The control will not have any support provided.

INTERVENTIONS:
Behavioral: HOPE Intervention — Participants used the Health Checkins Platform for 12 weeks for emotional support and to obtain pain management tools
  Arms: HOPE Intervention

SUMMARY:
The investigators have created an online peer support platform for chronic pain patients on opioid medications. This platform provides peer support and online mental health counselor run support groups to help participants manage pain and not abuse opioid medications.

DETAILED DESCRIPTION:
This study determined the feasibility, acceptability, and preliminary efficacy of an online support and risk reduction platform to prevent opioid misuse and abuse. This is an urgent area of research; opioid misuse/abuse has reached epidemic proportions in recent years. It is linked to causing the largest drug epidemic in the history of the United States and has become the top priority of the US Surgeon General. Because the opioid crisis (including heroin use) is believed to have largely originated from chronic pain patients' opioid prescriptions, this application will initially focus on the needs of chronic pain patients on opioids who are high risk for addiction and overdose. Later versions of the technology will expand to the broader population of people affected by the opioid crisis, including heroin users.

Although low cost, novel interventions are needed to reduce opioid misuse and abuse, before they lead to addiction and fatal overdose, only 6 behavioral (non-pharmacological) randomized controlled trials have been successfully conducted in this area to date (with our group having conducted one of them), creating a tremendous need for solutions to the opioid crisis. Building off extensive preliminary research that our team conducted, including piloting technology-based behavior change interventions among chronic pain patients, and developing artificial intelligence (AI)-based prediction models of opioid outcomes, we propose to design and test the feasibility, acceptability, and preliminary efficacy of an online peer social support and clinical counseling community to reduce opioid misuse/abuse among chronic pain sufferers.

ELIGIBILITY:
Inclusion Criteria: adults over 18, COMM scores at risk of misuse, prescribed opioids by doctor -

Exclusion Criteria: cancer patients, elicit drug users, under 18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder scale 7 scores | 12 weeks
  Anxiety levels

SECONDARY OUTCOMES:
Beck Depression Inventory scores | 12 weeks
  Depression levels
Current Opioid Misuse Measure scores | 12 weeks
  common opioid misuse measure

CONTACTS AND LOCATIONS:
Locations (1):
- ElevateU, Corona del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No